CLINICAL TRIAL: NCT01795300
Title: Randomized Comparison of Proton and Carbon Ion Radiotherapy With Advanced Photon Radiotherapy in Skull Base Meningiomas: The PINOCCHIO Trial.
Brief Title: Comparison of Proton and Carbon Ion Radiotherapy With Advanced Photon Radiotherapy in Skull Base Meningiomas: The PINOCCHIO Trial.
Acronym: PINOCCHIO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Organizational reasons
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PINOCCHIO
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Skull Base Meningioma
MeSH Terms: interventions — Heavy Ion Radiotherapy; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Carbon Ion Radiotherapy (Experimental): Treatment Schedule Carbon Ion Radiation Total Dose 45 Gy E, 15 fractions, 3 Gy E single dose
  Interventions: Radiation: Carbon Ion Radiotherapy
- Proton Therapy (Experimental): Treatment Schedule Proton Radiation Total Dose 45 Gy E, 15 fractions, 3 Gy E single dose
  Interventions: Radiation: Proton Therapy
- Hypofractionated Photon Therapy (Experimental): Treatment Schedule Photon Radiation 3 Gy E Total Dose 45 Gy E, 15 fractions, 3 Gy E single dose
  Interventions: Radiation: Hypofractionated Photon Radiotherapy
- Conventional Photon Radiotherapy (Active Comparator): Treatment Schedule Photon Radiation 1.8 Gy E Total Dose 57.6 Gy Gy E, 32 fractions, 1.8 Gy E single dose
  Interventions: Radiation: Conventional Photon Radiotherapy

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy — Patients will be immobilized using an individually manufactured head mask for treatment planning and RT. Contrast-enhanced CT as well as MR-imaging will be performed for target volume definition. OAR such as the brain stem, optic nerves, chiasm and spinal chord will be contoured. The fractionation scheme will be taken into account for dose prescription, as well as DVH-characteristics and clinical parameters of the invidivual patient.
  The Gross Tumor Volume (GTV) will be defined as the contrast-enhancing lesion on MRI on T1-weighted MR-imaging. Amino-Acid-PET or DOTATOC-PET may be used in addition to contrast-enhanced MRI for target volume definition but is not mandatory.The Clinical Target Volume (CTV) will be defined adding 1-2mm safety margin to the GTV.
  Arms: Carbon Ion Radiotherapy
Radiation: Proton Therapy — As described previously, patients will be immobilized using an individually manufactured head mask for treatment planning and RT. Contrast-enhanced CT as well as MR-imaging will be performed for target volume definition. OAR such as the brain stem, optic nerves, chiasm and spinal chord will be contoured. Dose constraints of normal tissue will be respected according to Emami et al. (33). The fractionation scheme will be taken into account for dose prescription, as well as DVH-characteristics and clinical parameters of the invidivual patient.
  The Gross Tumor Volume (GTV) will be defined as the contrast-enhancing lesion on MRI on T1-weighted MR-imaging. Amino-Acid-PET or DOTATOC-PET may be used in addition to contrast-enhanced MRI for target volume definition but is not mandatory.The Clinical Target Volume (CTV) will be defined adding 1-2mm safety margin to the GTV.
  Arms: Proton Therapy
Radiation: Hypofractionated Photon Radiotherapy — Treatment Planning for Photon Radiotherapy will be performed using the Planning Systems available at the Department of Radiation Oncology in Heidelberg, Germany (including Masterplan/Nucletron, Virtuos-Konrad/Siemens, or Precisis/STP/Stryker-Leibinger, or the Tomotherapy Software). Carbon ion and proton RT planning is performed using the treatment planning software PT-Planning (Siemens, Erlangen, Germany) including biologic plan optimization. Biologically effective dose distributions will be calculated using the a/ß ratio for meningioma as well as for the endpoint late toxicity to the brain. Patient positioning prior to radiotherapy will be evaluated by comparison of x-rays to the DRRs. Set up deviations >3mm are corrected prior to radiotherapy.
  To the target volume defined for photon treatment, a total dose of 52.2 Gy E - 57.6 Gy E is applied in single fractions of 1.8Gy E. In the 3Gy E Photon arm, photon radiotherapy will be delivered to a total dose of 45 Gy E in 15 fractions.
  Arms: Hypofractionated Photon Therapy
Radiation: Conventional Photon Radiotherapy — Treatment Planning for Photon Radiotherapy will be performed using the Planning Systems available at the Department of Radiation Oncology in Heidelberg, Germany (including Masterplan/Nucletron, Virtuos-Konrad/Siemens, or Precisis/STP/Stryker-Leibinger, or the Tomotherapy Software). Carbon ion and proton RT planning is performed using the treatment planning software PT-Planning (Siemens, Erlangen, Germany) including biologic plan optimization. Biologically effective dose distributions will be calculated using the a/ß ratio for meningioma as well as for the endpoint late toxicity to the brain. Patient positioning prior to radiotherapy will be evaluated by comparison of x-rays to the DRRs. Set up deviations >3mm are corrected prior to radiotherapy.
  Arms: Conventional Photon Radiotherapy

SUMMARY:
In PINOCCHIO-Triayl, carbon ion radiotherapy is compared to proton and advanced photon radiotherapy in patients with skull base meningiomas. There will be two treatment arms with photons, one arm with hypofractionated photon radiotherapy, and one arm with conventional fractionation. The study is designed as descriptive study on feasibility of the investigated therapies aiming at a comparison of toxicities. The study will serve as a basis for further larger randomized protocols comparing efficacy of the therapies, assuming toxicity is comparable in all four treatment arms. Primary endpoint is toxicity, secondary endpoints are overall survival, progression-free survival and quality of life.

ELIGIBILITY:
Inclusion Criteria

Patients meeting all of the following criteria will be considered for admission to the trial:

* Histologically or imaging confirmed skull base meningioma
* macroscopic tumor - Simpson Grade 4 or 5
* age ≥ 18 years of age
* Karnofsky Performance Score >=60
* For women with childbearing potential, (and men) adequate contraception (sexual abstinence, estrogen- or gestagen containing contraceptive medication etc.)
* Female participants: No pregnancy present (pregnancy test required)
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion criteria:

Patients presenting with any of the following criteria will not be included in the trial:

* refusal of the patients to take part in the study
* previous radiotherapy of the brain
* histologically confirmed atypical or anaplastic meningioma
* optic nerve sheath meningioma (ONSM)
* Patients who have not yet recovered from acute toxicities of prior therapies
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Toxicity graded according to CTCAE Version 4.1 after 1 year | 1 year
  Toxicity graded according to CTCAE Version 4.1 after 1 year

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival
Progression-free survival | 3 years
  Progression-free survival
Quality of Life | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany